CLINICAL TRIAL: NCT02829437
Title: Endometrial Stromal Tumors: an Observational Study
Brief Title: Observational Study on Endometrial Stromal Tumors
Acronym: EST
Status: Recruiting | Type: Observational
Sponsor: Italian Sarcoma Group (Network)
Responsible Party: Sponsor
Other Study IDs: ISG EST
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Endometrial Stromal Tumors
MeSH Terms: conditions — Endometrial Stromal Tumors | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Paraffin-embedded pathologic tissue used for diagnostic confirmation purposes only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Retrospective Observational Group: Patients who received treatment for EST Patients with EST diagnosis prior August 2016
  Interventions: Other: Treatment for EST
- Prospective Observational Group: Patients who will receive treatment for EST Patients with EST diagnosis after August 2016
  Interventions: Other: Treatment for EST

INTERVENTIONS:
Other: Treatment for EST — Surgery and/or Chemotherapy and or/radiotherapy for EST treatment according to disease guidelines: no specific treatment is imposed by protocol (observational study)

SUMMARY:
Observational, retrospective and prospective study on Endometrial Stromal Tumor (EST)

DETAILED DESCRIPTION:
Observational, retrospective and prospective study on EST aimed to understand more about its biology, natural history and antitumor activity of different treatment options.

This study will collect data in prospective and retrospective way of patients affected by EST and treated according disease guidelines and local practices.

The study will also review the diagnosis by a central expert pathologist in order to its confirmation

ELIGIBILITY:
Inclusion Criteria:

* patients with a diagnosis of Endometrial Stromal Tumor (EST) according to the World Health Organization (WHO) classification 2003 or 2014
* Informed consent signature

Exclusion Criteria:

* patients with different diagnosis from EST

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients with a diagnosis of Endometrial Stromal Tumor (EST)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-10; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Disease natural history | Through survival, an average of 5 years
  Collection of data on the natural history of endometrial stromal tumors

SECONDARY OUTCOMES:
Disease diagnosis and classification | At the time of diagnosis, an average of 1 month
  Highlight some main issues in pathologic diagnosis of these tumors and their classification
Chemotherapy received treatment | Through treatment completion, an average of 24 month
  Number and type of chemotherapy agents received for EST treatment

CONTACTS AND LOCATIONS:
Overall Officials: Paolo G Casali, MD, Study Chair — Italian Sarcoma Group
Locations (13):
- Italy (13):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori - IRST, Meldola, FC
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, MI
  - Istituto Europeo di Oncologia, Milan, MI
  - Azienda Ospedaliera Universitaria Paolo Giaccone, Palermo, PA
  - Centro di Riferimento Oncologico di Aviano, Aviano, PD
  - Istituto Oncologico Veneto, Padua, PD
  - Fondazione del Piemonte per l'Oncologia IRCC Candiolo, Candiolo, Torino
  - Policlinico S.Orsola Malpighi - Unit of Medical Oncology, Bologna
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Ospedale Misericordia e Dolce Ist. Toscano Tumori, Az. USL4, Prato
  - Campus Biomedico, Roma
  - Istituti Fisioterapici Ospitalieri di Roma, Roma

IPD SHARING:
Plan to Share IPD: Yes
Aggregate anonymized results will be available upon request at the end of the study

REFERENCES:
- [Background] Brooks SE, Zhan M, Cote T, Baquet CR. Surveillance, epidemiology, and end results analysis of 2677 cases of uterine sarcoma 1989-1999. Gynecol Oncol. 2004 Apr;93(1):204-8. doi: 10.1016/j.ygyno.2003.12.029. PMID 15047237
- [Background] Toro JR, Travis LB, Wu HJ, Zhu K, Fletcher CD, Devesa SS. Incidence patterns of soft tissue sarcomas, regardless of primary site, in the surveillance, epidemiology and end results program, 1978-2001: An analysis of 26,758 cases. Int J Cancer. 2006 Dec 15;119(12):2922-30. doi: 10.1002/ijc.22239. PMID 17013893
- [Background] Ali RH, Rouzbahman M. Endometrial stromal tumours revisited: an update based on the 2014 WHO classification. J Clin Pathol. 2015 May;68(5):325-32. doi: 10.1136/jclinpath-2014-202829. Epub 2015 Jan 16. PMID 25595274
- [Background] Tavassoli FA, Norris HJ. Mesenchymal tumours of the uterus. VII. A clinicopathological study of 60 endometrial stromal nodules. Histopathology. 1981 Jan;5(1):1-10. doi: 10.1111/j.1365-2559.1981.tb01761.x. PMID 7216172
- [Background] Dionigi A, Oliva E, Clement PB, Young RH. Endometrial stromal nodules and endometrial stromal tumors with limited infiltration: a clinicopathologic study of 50 cases. Am J Surg Pathol. 2002 May;26(5):567-81. doi: 10.1097/00000478-200205000-00003. PMID 11979087
- [Background] Su TF, Chao TK, Lee HS, Perng CL, Nieh S. Malignant potential of endometrial stromal tumor with limited infiltration: a case report. Int J Surg Pathol. 2014 Sep;22(6):559-63. doi: 10.1177/1066896913506934. Epub 2013 Oct 23. PMID 24155223
- [Background] Dong R, Pang Y, Mao H, Yang N, Liu P. Successful pregnancy following conservative management of low-grade endometrial stromal sarcoma: A case report. Oncol Lett. 2014 Apr;7(4):1039-1042. doi: 10.3892/ol.2014.1858. Epub 2014 Feb 7. PMID 24944665
- [Background] Choi MC, Kim G, Hwang YY. Fertility-sparing management combined with photodynamic therapy for endometrial stromal sarcoma: a case report. Photodiagnosis Photodyn Ther. 2014 Dec;11(4):533-6. doi: 10.1016/j.pdpdt.2014.07.007. Epub 2014 Aug 11. PMID 25125393
- [Background] Della Badia C, Karini H. Endometrial stromal sarcoma diagnosed after uterine morcellation in laparoscopic supracervical hysterectomy. J Minim Invasive Gynecol. 2010 Nov-Dec;17(6):791-3. doi: 10.1016/j.jmig.2010.07.001. PMID 20955991
- [Background] Park JY, Kim DY, Kim JH, Kim YM, Kim YT, Nam JH. The impact of tumor morcellation during surgery on the outcomes of patients with apparently early low-grade endometrial stromal sarcoma of the uterus. Ann Surg Oncol. 2011 Nov;18(12):3453-61. doi: 10.1245/s10434-011-1751-y. Epub 2011 May 4. PMID 21541824
- [Background] Shah JP, Bryant CS, Kumar S, Ali-Fehmi R, Malone JM Jr, Morris RT. Lymphadenectomy and ovarian preservation in low-grade endometrial stromal sarcoma. Obstet Gynecol. 2008 Nov;112(5):1102-8. doi: 10.1097/AOG.0b013e31818aa89a. PMID 18978112
- [Background] Dos Santos LA, Garg K, Diaz JP, Soslow RA, Hensley ML, Alektiar KM, Barakat RR, Leitao MM Jr. Incidence of lymph node and adnexal metastasis in endometrial stromal sarcoma. Gynecol Oncol. 2011 May 1;121(2):319-22. doi: 10.1016/j.ygyno.2010.12.363. Epub 2011 Jan 26. PMID 21276609
- [Background] Amant F, De Knijf A, Van Calster B, Leunen K, Neven P, Berteloot P, Vergote I, Van Huffel S, Moerman P. Clinical study investigating the role of lymphadenectomy, surgical castration and adjuvant hormonal treatment in endometrial stromal sarcoma. Br J Cancer. 2007 Nov 5;97(9):1194-9. doi: 10.1038/sj.bjc.6603986. Epub 2007 Sep 25. PMID 17895898
- [Background] Amant F, Coosemans A, Debiec-Rychter M, Timmerman D, Vergote I. Clinical management of uterine sarcomas. Lancet Oncol. 2009 Dec;10(12):1188-98. doi: 10.1016/S1470-2045(09)70226-8. PMID 19959075
- [Background] Rauh-Hain JA, del Carmen MG. Endometrial stromal sarcoma: a systematic review. Obstet Gynecol. 2013 Sep;122(3):676-83. doi: 10.1097/AOG.0b013e3182a189ac. PMID 23921879
- [Background] Gadducci A, Sartori E, Landoni F, Zola P, Maggino T, Urgesi A, Lissoni A, Losa G, Fanucchi A. Endometrial stromal sarcoma: analysis of treatment failures and survival. Gynecol Oncol. 1996 Nov;63(2):247-53. doi: 10.1006/gyno.1996.0314. PMID 8910635
- [Background] Chu MC, Mor G, Lim C, Zheng W, Parkash V, Schwartz PE. Low-grade endometrial stromal sarcoma: hormonal aspects. Gynecol Oncol. 2003 Jul;90(1):170-6. doi: 10.1016/s0090-8258(03)00258-0. PMID 12821359
- [Background] Li AJ, Giuntoli RL 2nd, Drake R, Byun SY, Rojas F, Barbuto D, Klipfel N, Edmonds P, Miller DS, Karlan BY. Ovarian preservation in stage I low-grade endometrial stromal sarcomas. Obstet Gynecol. 2005 Dec;106(6):1304-8. doi: 10.1097/01.AOG.0000185511.91694.1e. PMID 16319256
- [Background] Kim WY, Lee JW, Choi CH, Kang H, Kim TJ, Kim BG, Lee JH, Bae DS. Low-grade endometrial stromal sarcoma: a single center's experience with 22 cases. Int J Gynecol Cancer. 2008 Sep-Oct;18(5):1084-9. doi: 10.1111/j.1525-1438.2007.01159.x. Epub 2007 Dec 27. PMID 18179547
- [Background] Altman AD, Nelson GS, Chu P, Nation J, Ghatage P. Uterine sarcoma and aromatase inhibitors: Tom Baker Cancer Centre experience and review of the literature. Int J Gynecol Cancer. 2012 Jul;22(6):1006-12. doi: 10.1097/IGC.0b013e31825b7de8. PMID 22740004
- [Background] Leath CA 3rd, Huh WK, Hyde J Jr, Cohn DE, Resnick KE, Taylor NP, Powell MA, Mutch DG, Bradley WH, Geller MA, Argenta PA, Gold MA. A multi-institutional review of outcomes of endometrial stromal sarcoma. Gynecol Oncol. 2007 Jun;105(3):630-4. doi: 10.1016/j.ygyno.2007.01.031. Epub 2007 Feb 23. PMID 17320937
- [Background] Thomas MB, Keeney GL, Podratz KC, Dowdy SC. Endometrial stromal sarcoma: treatment and patterns of recurrence. Int J Gynecol Cancer. 2009 Feb;19(2):253-6. doi: 10.1111/IGC.0b013e3181999c5f. PMID 19396004
- [Background] Omura GA, Major FJ, Blessing JA, Sedlacek TV, Thigpen JT, Creasman WT, Zaino RJ. A randomized study of adriamycin with and without dimethyl triazenoimidazole carboxamide in advanced uterine sarcomas. Cancer. 1983 Aug 15;52(4):626-32. doi: 10.1002/1097-0142(19830815)52:43.0.co;2-e. PMID 6344983
- [Background] Cheng X, Yang G, Schmeler KM, Coleman RL, Tu X, Liu J, Kavanagh JJ. Recurrence patterns and prognosis of endometrial stromal sarcoma and the potential of tyrosine kinase-inhibiting therapy. Gynecol Oncol. 2011 May 1;121(2):323-7. doi: 10.1016/j.ygyno.2010.12.360. Epub 2011 Jan 28. PMID 21277011
- [Background] Piver MS, Rutledge FN, Copeland L, Webster K, Blumenson L, Suh O. Uterine endolymphatic stromal myosis: a collaborative study. Obstet Gynecol. 1984 Aug;64(2):173-8. PMID 6738952
- [Background] Sutton G, Blessing JA, Park R, DiSaia PJ, Rosenshein N. Ifosfamide treatment of recurrent or metastatic endometrial stromal sarcomas previously unexposed to chemotherapy: a study of the Gynecologic Oncology Group. Obstet Gynecol. 1996 May;87(5 Pt 1):747-50. doi: 10.1016/0029-7844(96)00003-8. PMID 8677079